CLINICAL TRIAL: NCT04147286
Title: Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Safety and Efficacy of Atorvastatin to Reduce Inflammation After Tuberculosis Treatment Completion in HIV-infected and HIV-uninfected Adults Measured by FDG-PET/CT
Brief Title: Atorvastatin to Reduce Inflammation After Tuberculosis Treatment Completion
Acronym: StatinTB
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Zurich (Other); University of Namibia (Other); University of Bern (Other); University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Prof Friedrich Thienemann, Associate Professor and research group leader, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC 675/2019; RIA2017T-2004 (Other Grant/Funding Number: EDCTP); HREC 675/2019 (Other: IRB (University of Cape Town))
Record Dates: First submitted 2019-10-23; First posted 2019-11-01 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis, Pulmonary
Keywords: tuberculosis; HIV; COPD; inflammation
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis; Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: This is a proof-of-concept phase IIB, double-blind, randomized, placebo-controlled trial to evaluate the safety and efficacy of 40 mg atorvastatin to reduce persistent lung inflammation after successful TB treatment completion in HIV-infected and HIV-uninfected adults measured by PET/CT.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, randomized, placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Arm B) (Active Comparator): 12 weeks of 40 mg atorvastatin therapy per os daily
  Interventions: Drug: Atorvastatin 40mg
- Placebo (Arm C) (Placebo Comparator): Identical placebo tablet is taken per os daily
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Atorvastatin 40mg — 12 weeks of 40 mg atorvastatin therapy per os
  Arms: Atorvastatin (Arm B)
Drug: Placebo oral tablet — Identical placebo
  Arms: Placebo (Arm C)

SUMMARY:
This is a proof-of-concept phase IIB, double-blind, randomized, placebo-controlled trial to evaluate the safety and efficacy of 40 mg atorvastatin to reduce persistent lung inflammation after successful TB treatment completion in HIV-infected and HIV-uninfected adults measured by PET/CT.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (Mtb) causes 1.8 million deaths annually. Sub-Saharan Africa carries the highest burden of tuberculosis (TB) with recurrent TB rates between 3-5% after treatment completion accounting for 10-30% of all cases within some TB control programs. Multiple risk factors have been identified to cause recurrent diseases. A recent study has identified persistent lesion activity by 18F-fluoro-D-glucose positron emission tomography (PET/CT) suggesting ongoing inflammation and Mtb mRNA suggesting ongoing infection after cure. The presence of inflammation and mRNA implies that current curative treatment options for pulmonary TB may not eradicate Mtb in most patients and more potent treatment options including host-directed therapy (HDT) to sterilize during or after TB treatment is required.

Mtb accumulates host cholesterol ester in foamy macrophages and utilizes cholesterol for its persistence within macrophages. Statins lower cholesterol in cardiovascular diseases through inhibition of HMG-CoA reductase, the rate-controlling enzyme of the mevalonate pathway. In addition, statins also have broad-range immune-modulatory and anti-inflammatory properties.

As previously reported in pre-clinical models that statins reduced Mtb burden by enhancing autophagy, phagosomal maturation and decreasing pulmonary pathology, suggesting a role for statins as HDT in TB. Others reported that statins as adjunctive therapy reduced the time for TB cure and decreased lung pathology in mice. A recent population-based study consisting of 1 million people reported that statin treatment was associated with a decreased risk of active TB.

This protocol builds upon successful studies suggesting that directly monitoring lung pathology using PET/CT correlates better with treatment outcome than culture and persistent inflammation measured by PET/CT is present after tuberculosis cure in most patients.

The investigators propose a proof-of-concept phase IIB, double-blind, randomized, placebo-controlled trial to evaluate the safety and efficacy of 40 mg atorvastatin per os daily to reduce persistent inflammation after TB treatment completion in HIV-infected and HIV-uninfected adults measured by PET/CT.

If successful, this trial has proven that statins as HDT can be safe and effective adjunctive therapy to TB treatment in general and further efficacy trials can be undertaken to translate the results of this trial into reduced TB relapse rate and reduced post-TB chronic lung disease, thus decreased long-term TB-related morbidity.

The investigators hypothesize that 12 weeks of 40 mg atorvastatin therapy per os initiated at the end of successful TB treatment in HIV infected and HIV-uninfected participants will significantly reduce persistent lung inflammation on PET/CT scan.

Primary objective To compare persistent lung inflammation measured by total lung glycolysis (TLG) on PET/CT after 12 weeks of 40 mg atorvastatin therapy and placebo.

ELIGIBILITY:
Inclusion Criteria

1. Has completed the written informed consent process prior to undergoing any pre-screening or screening evaluations and willing to undergo HIV testing
2. Age 18 to 65 years with body weight from 50 kg to 90 kg
3. Clinical response to TB treatment and sputum culture negative at week 16
4. Completed a 24-week course of standard TB treatment (4RHZE/2RH)
5. Defined as "cured" by the TB Control Program of South Africa

   Laboratory parameters within 30 days before enrolment:
6. For HIV-infected participants: receiving antiretroviral therapy for at least 12 weeks and suppressed HIV viral load within 30 days prior to enrolment
7. For HIV-infected participants: CD4 counts above 350 cells/µL within 30 days prior to enrolment
8. AST and ALT <3x upper limit of normal (ULN)
9. Creatinine <2x ULN
10. Hemoglobin >7.0 g/dL
11. Platelet count >50 x109 cells/L
12. Creatinine kinase <2x ULN
13. Able and willing to return to follow-up
14. Willing to have samples, including DNA, stored
15. Willing to consistently practice a highly reliable method of pregnancy prevention

Exclusion criteria

1. Acute illness
2. Fever (temperature >38.0 degrees centigrade)
3. Participant receiving any type of lipid lowering agent at the time of screening, within three months prior to screening or likely to require any lipid lowering agent in the near future.
4. Known allergy or contraindications to the investigational drug or any other statins
5. Evidence of drug-resistant TB
6. Extrapulmonary TB, including pleural TB and/or large pleural effusion
7. Pregnant or desiring/trying to become pregnant in the next 6 months
8. Unable to take oral medications
9. Diabetes as defined by point of care HbA1c≥6.5, random glucose≥200mg/dL (or 11.1mmol/L), fasting plasma glucose≥126mg/dL (or 7.0mmol/L), or the presence of any anti-diabetic agent (including traditional medicines) as a concomitant medicine
10. Disease complications or concomitant illnesses that may compromise safety or interpretation of trial endpoints, such as known diagnosis of chronic inflammatory condition (e.g. sarcoidosis, rheumatoid arthritis, connective tissue disorder)
11. Use of immunosuppressive medications, such as TNF-alpha inhibitors or systemic or inhaled corticosteroids, within the past 2 weeks
12. Use of any investigational drug in the previous 3 months
13. Alcohol and substance abuse which might interfere with medication adherence during the trial
14. Any person for whom the physician feels this study is not appropriate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Total lung glycolysis (TLG) on PET/CT imaging | 12 weeks
  The primary outcome measure is total lung glycolysis (TLG) on PET/CT imaging.
  Total lung glycolysis (TLG), is the total glycolytic activity (TGA) in regions of interest (both lungs). Primary outcome measurement is semi-automated using nuclear medicine medical imaging software (MIM Software Inc.). Total lung masks are drawn on every participant's PET/CT scans. Glycolytic activity is derived for each lung (SUVbw*mL), total lung glycolytic activity is the sum of both lungs TGA.

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Thienemann, MD, Principal Investigator — University of Cape Town; Reto Guler, PhD, Study Chair — University of Cape Town
Locations (1):
- General Medicine & Global Health, Cape Heart Institute, Faculty of Health Sciences, University of Cape Town, Observatory, WC, South Africa